CLINICAL TRIAL: NCT06897722
Title: Psoriasis and Periodontitis Are Chronic Inflammatory Diseases Characterized by Immune Dysregulation and Systemic Inflammatory Burden. Both Conditions Share Key Inflammatory Mediators, Including Tumor Necrosis Factor-alpha (TNF-α), Interleukin-17A (IL-17A), and YKL-40, Which Contribute to Tissue Destruction and Disease Progression. This Study Aimed to Investigate the Association Between Psoriasis and Periodontal Diseases by Evaluating Clinical Periodontal Parameters and Measuring TNF-α, IL-17A, and YKL-40 Levels in Gingival Crevicular Fluid (GCF) and Serum.
Brief Title: Evaluation of TNF-α, IL-17A, and YKL-40 in GCF and Serum of Psoriasis Patients and Healthy Controls
Status: Active, not recruiting | Type: Observational
Sponsor: Zhala Vatankha Sain (Other)
Responsible Party: Sponsor-Investigator, Zhala Vatankha Sain, Researcher, Department of Periodontology, Akdeniz University, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: AkdenizU Organization
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-11

CONDITIONS: Psoriasis (PsO); Periodontal Disease
Keywords: Psoriasis; Periodontitis; GCF; TNF-α; IL-17A; YKL-40; Serum Markers
MeSH Terms: conditions — Psoriasis; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- 1 group : Control (C): 1 group : Control (C): Healthy individuals without psoriasis, gingivitis or periodontitis.
  Interventions: Diagnostic Test: TNF-α analysis in GCF; Diagnostic Test: IL-17A analysis in GCF; Diagnostic Test: YKL-40 analysis in GCF; Diagnostic Test: TNF-α analysis in Serum; Diagnostic Test: İL-17A analysis in Serum; Diagnostic Test: YKL-40 analysis in Serum; Diagnostic Test: Periodontal assesment
- 2. group Gingivitis (G): Gingivitis (G): Individuals diagnosed with gingivitis but without psoriasis.
  Interventions: Diagnostic Test: TNF-α analysis in GCF; Diagnostic Test: IL-17A analysis in GCF; Diagnostic Test: YKL-40 analysis in GCF; Diagnostic Test: TNF-α analysis in Serum; Diagnostic Test: İL-17A analysis in Serum; Diagnostic Test: YKL-40 analysis in Serum; Diagnostic Test: Periodontal assesment
- 3. group Periodontitis (P): 3. group Periodontitis (P): Individuals diagnosed with periodontitis but without psoriasis.
  Interventions: Diagnostic Test: TNF-α analysis in GCF; Diagnostic Test: IL-17A analysis in GCF; Diagnostic Test: YKL-40 analysis in GCF; Diagnostic Test: TNF-α analysis in Serum; Diagnostic Test: İL-17A analysis in Serum; Diagnostic Test: YKL-40 analysis in Serum; Diagnostic Test: Periodontal assesment
- 4. group Psoriasis with gingivitis (PS+G): 4. group Psoriasis with gingivitis (PS+G): Individuals diagnosed with gingivitis and psoriasis.
  Interventions: Diagnostic Test: TNF-α analysis in GCF; Diagnostic Test: IL-17A analysis in GCF; Diagnostic Test: YKL-40 analysis in GCF; Diagnostic Test: TNF-α analysis in Serum; Diagnostic Test: İL-17A analysis in Serum; Diagnostic Test: YKL-40 analysis in Serum; Diagnostic Test: Periodontal assesment
- 5. group Psoriasis with Periodontitis (PS+P): 5. group Psoriasis with Periodontitis (PS+P): Individuals diagnosed with psoriasis and periodontitis.
  Interventions: Diagnostic Test: TNF-α analysis in GCF; Diagnostic Test: IL-17A analysis in GCF; Diagnostic Test: YKL-40 analysis in GCF; Diagnostic Test: TNF-α analysis in Serum; Diagnostic Test: İL-17A analysis in Serum; Diagnostic Test: YKL-40 analysis in Serum; Diagnostic Test: Periodontal assesment

INTERVENTIONS:
Diagnostic Test: TNF-α analysis in GCF — The primary intervention will involve the non-invasive collection of GCF samples using Periopaper strips. The strips will be placed into the gingival sulcus for 30 seconds and then stored at -80°C until analysis. The analysis of TNF-α levels in gingival crevicular fluid (GCF) will be performed using ELISA.
Diagnostic Test: IL-17A analysis in GCF — The primary intervention involves the non-invasive collection of GCF samples using periopaper strips. Periopaper strips are placed into the gingival sulcus for 30 seconds, then stored at -80°C until analysis. Analysis of TNF-α levels in gingival crevicular fluid (GCF) will be performed using ELISA.
Diagnostic Test: YKL-40 analysis in GCF — The primary intervention involves the non-invasive collection of GCF samples using periopaper strips. Periopaper strips are placed into the gingival sulcus for 30 seconds, then stored at -80°C until analysis. Analysis of TNF-α levels in gingival crevicular fluid (GCF) will be performed using ELISA.
Diagnostic Test: TNF-α analysis in Serum — The intervention will involve venous blood collection for serum analysis. Venous blood will be drawn, allowed to clot, will be centrifuged at 3,000 rpm for 10 minutes, and will be stored at -80°C until analysis.
Diagnostic Test: İL-17A analysis in Serum — The intervention will involve venous blood collection for serum analysis. Venous blood will be drawn, allowed to clot, will be centrifuged at 3,000 rpm for 10 minutes, and will be stored at -80°C until analysis.
Diagnostic Test: YKL-40 analysis in Serum — The intervention will involve venous blood collection for serum analysis. Venous blood will be drawn, allowed to clot, will be centrifuged at 3,000 rpm for 10 minutes, and will be stored at -80°C until analysis.
Diagnostic Test: Periodontal assesment — Comprehensive periodontal assessments will be conducted, including Plaque Index (PI), Bleeding on Probing (BOP), Probing Pocket Depth (PPD), and Clinical Attachment Level (CAL).

SUMMARY:
Background:

Psoriasis is a chronic inflammatory skin disease that affects 2-3% of the global population and is linked to immune dysregulation and systemic inflammation. Periodontitis, a chronic inflammatory gum disease, leads to the destruction of gum tissues and bone. Both conditions share common inflammatory pathways, with key immune mediators such as tumor necrosis factor-alpha (TNF-α), interleukin-17A (IL-17A), and YKL-40 playing a role in tissue destruction and disease progression. However, the biological mechanisms linking psoriasis and periodontitis remain unclear, and few studies have examined localized inflammatory responses in the gums of psoriasis patients.

Objectives and Methods:

This study aims to evaluate the relationship between psoriasis and periodontitis by measuring TNF-α, IL-17A, and YKL-40 levels in both gingival crevicular fluid (GCF) and serum. A total of 100 participants will be recruited and categorized into three groups:

Control (C): Healthy individuals without psoriasis or periodontitis. Gingivitis (G): Individuals diagnosed with gingivitis but without psoriasis. Periodontitis (P): Individuals diagnosed with periodontitis but without psoriasis.

Psoriasis with gingivitis (PS+G): Individuals diagnosed with gingivitis but without psoriasis.

Psoriasis with Periodontitis (PS+P): Individuals with both psoriasis and periodontitis.

All participants will undergo periodontal examinations, including plaque index (PI), bleeding on probing (BOP), probing pocket depth (PPD), and clinical attachment level (CAL). GCF and blood samples will be collected, and biomarker levels will be analyzed using enzyme-linked immunosorbent assay (ELISA).

Expected Outcomes and Clinical Relevance:

The study will investigate whether systemic inflammation in psoriasis contributes to periodontal disease progression. If psoriasis patients show higher inflammatory biomarker levels, it may suggest a shared immunopathogenic mechanism.

The results may contribute to:

Early detection strategies for periodontitis in psoriasis patients. Targeted anti-inflammatory therapies for both conditions. Interdisciplinary collaboration between dermatologists and periodontists for better management.

This study is the first to evaluate TNF-α and YKL-40 in the GCF of psoriasis patients, filling a critical gap in the literature regarding localized immune responses. The results could also help identify potential biomarkers that may be useful for monitoring disease progression and treatment responses in psoriasis and periodontitis patients.

Conclusion:

By investigating the inflammatory relationship between psoriasis and periodontitis, this study aims to uncover new insights into the immune system's role in chronic inflammatory diseases. Understanding these mechanisms could lead to improved diagnostic tools, prevention strategies, and personalized treatment approaches for patients affected by both conditions.

DETAILED DESCRIPTION:
Psoriasis and periodontitis are chronic inflammatory diseases that share key immunopathological mechanisms. Psoriasis is primarily a dermatological condition, but it also exhibits systemic inflammatory characteristics that may contribute to comorbidities such as periodontitis. Periodontitis, a chronic immune-inflammatory condition of the supporting structures of the teeth, is similarly characterized by sustained inflammatory responses and tissue destruction.

Emerging evidence suggests that these two diseases may be biologically linked through shared inflammatory pathways. Among the common mediators, tumor necrosis factor-alpha (TNF-α), interleukin-17A (IL-17A), and YKL-40 play prominent roles in the pathogenesis of both conditions. TNF-α contributes to immune activation, tissue breakdown, and bone resorption. IL-17A, associated with Th17-mediated responses, promotes keratinocyte proliferation and inflammatory cell infiltration in psoriasis, while driving extracellular matrix degradation and osteoclastogenesis in periodontitis. YKL-40, a glycoprotein involved in tissue remodeling and inflammation, has been proposed as a potential biomarker for chronic inflammatory diseases, including psoriasis and periodontitis.

While elevated levels of these markers have been individually observed in serum or tissues of patients with either condition, limited data exist on their expression in both systemic and local environments-particularly within the gingival crevicular fluid (GCF) of psoriasis patients. This study will address this gap by assessing TNF-α, IL-17A, and YKL-40 levels in GCF and serum samples of individuals with and without psoriasis and periodontal disease.

Through a cross-sectional, case-control study design, this research aims to investigate whether systemic inflammation associated with psoriasis correlates with increased periodontal inflammation and whether common biomarkers may indicate a shared pathogenic mechanism. Understanding this potential link could lead to improved interdisciplinary management strategies and earlier identification of periodontal risk in patients with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years.
2. Confirmed diagnosis of chronic plaque psoriasis (for PS+G, PS+P group) by a board-certified dermatologist.
3. Diagnosis of Gingivitis and Stage II or III, Grade B or C periodontitis (for P and PS+P groups) based on the 2017 World Workshop on the Classification of Periodontal Diseases and Conditions.
4. At least 20 remaining teeth.
5. No history of systemic conditions that could affect periodontal health, such as diabetes mellitus, autoimmune diseases, or cardiovascular diseases.
6. No prior periodontal treatment within the last 6 months.
7. No use of antibiotics, anti-inflammatory medications, or immunosuppressive drugs in the last 3 months.
8. Non-smokers or those who have not smoked in the past year.
9. Willingness to participate voluntarily and provide written informed consent.

Exclusion Criteria:

1. Age below 25 or above 65 years.
2. Diagnosis of any systemic inflammatory disease other than psoriasis, such as rheumatoid arthritis, inflammatory bowel disease, or systemic lupus erythematosus.
3. History of malignancy or chemotherapy/radiotherapy treatment.
4. Use of antibiotics, corticosteroids, or immunosuppressive drugs within the last 3 months.
5. Pregnant or lactating women.
6. Current smokers or individuals who have smoked within the last year.
7. History of substance abuse or chronic alcohol consumption.
8. Presence of acute infections, including oral or systemic infections.
9. Refusal to sign the informed consent form or inability to comply with the study protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes 100 participants from Akdeniz University, Turkey, categorized into five groups (n=20 each):
  Control (C): Healthy individuals without psoriasis or periodontitis, Gingivitis (G): Individuals diagnosed with gingivitis but without psoriasis, Periodontitis (P): Individuals with Stage II/III, Grade B/C periodontitis, but without psoriasis, Psoriasis with gingivitis (PS+G): Individuals diagnosed with gingivitis but without psoriasis, Psoriasis with Periodontitis (PS+P): Individuals with both psoriasis and periodontitis.
  Participants are 25-65 years old, non-smokers, with at least 20 teeth, and no systemic conditions affecting periodontal health. Psoriasis diagnoses are confirmed by a board-certified dermatologist; gingivitis and periodontitis is diagnosed per 2017 classification criteria.
  This study analyzes TNF-α, IL-17A, and YKL-40 levels in serum and gingival crevicular fluid (GCF) to explore the immunoinflammatory link between psoriasis and periodontitis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
TNF-α levels in gingival crevicular fluid (GCF) | At baseline (single visit)
  Levels of TNF-α will be measured using ELISA in GCF samples collected at baseline.
TNF-α levels in serum | At baseline (single visit).
  Levels of TNF-α will be measured using ELISA in serum samples collected at baseline.
IL-17A levels in gingival crevicular fluid (GCF) | At baseline (single visit).
  Levels of İL-17A will be measured using ELISA in serum samples collected at baseline.
IL-17A levels in serum | At baseline (single visit).
  Levels of IL-17A will be measured using ELISA in GCF samples collected at baseline.
YKL-40 levels in gingival crevicular fluid (GCF) | At baseline (single visit).
  Levels of YKL-40 will be measured using ELISA in GCF samples collected at baseline.
YKL-40 levels in serum | At baseline (single visit).
  Levels of TNF-α will be measured using ELISA in serum samples collected at baseline.
Periodontal assesment | At baseline (single visit)
  Probing Pocket Depth (PPD), Clinical Attachment Level (CAL), Bleeding on Probing (BOP), Plaque Index (PI) collected at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zhala Vatankha Sain, DDS, Principal Investigator — Akdeniz University, Faculty of Dentistry, Department of Periodontology; Kemal Üstün, Prof., Study Chair — Akdeniz University, Faculty of Dentistry, Department of Periodontology; Özlem Daltaban, Assoc. Prof., Study Director — Akdeniz University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Akdeniz University Faculty of Dentistry, Akdeniz University Hospital, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not been finalized. Future data-sharing plans will depend on institutional policies, ethical considerations, and applicable regulatory requirements.

REFERENCES:
- [Background] Kong Y, Zhang S, Su X, Peng D, Su Y. Serum levels of YKL-40 are increased in patients with psoriasis: a meta-analysis. Postgrad Med. 2019 Aug;131(6):405-412. doi: 10.1080/00325481.2019.1643634. Epub 2019 Jul 22. PMID 31298974
- [Background] Zhang X, Gu H, Xie S, Su Y. Periodontitis in patients with psoriasis: A systematic review and meta-analysis. Oral Dis. 2022 Jan;28(1):33-43. doi: 10.1111/odi.13617. Epub 2020 Sep 18. PMID 32852860
- [Background] Mendes VS, Cota LOM, Costa AA, Oliveira AMSD, Costa FO. Periodontitis as another comorbidity associated with psoriasis: A case-control study. J Periodontol. 2019 Apr;90(4):358-366. doi: 10.1002/JPER.18-0394. Epub 2018 Nov 28. PMID 30387155
- [Background] Armstrong AW, Puig L, Joshi A, Skup M, Williams D, Li J, Betts KA, Augustin M. Comparison of Biologics and Oral Treatments for Plaque Psoriasis: A Meta-analysis. JAMA Dermatol. 2020 Mar 1;156(3):258-269. doi: 10.1001/jamadermatol.2019.4029. PMID 32022825
- [Background] Marruganti C, Gaeta C, Falciani C, Cinotti E, Rubegni P, Alovisi M, Scotti N, Baldi A, Bellan C, Defraia C, Fiorino F, Valensin S, Bellini E, De Rosa A, D'Aiuto F, Grandini S. Are periodontitis and psoriasis associated? A pre-clinical murine model. J Clin Periodontol. 2024 Aug;51(8):1044-1053. doi: 10.1111/jcpe.13996. Epub 2024 May 3. PMID 38699834
- [Background] Gorska R, Gregorek H, Kowalski J, Laskus-Perendyk A, Syczewska M, Madalinski K. Relationship between clinical parameters and cytokine profiles in inflamed gingival tissue and serum samples from patients with chronic periodontitis. J Clin Periodontol. 2003 Dec;30(12):1046-52. doi: 10.1046/j.0303-6979.2003.00425.x. PMID 15002890
- [Background] Jimenez C, Carvajal D, Hernandez M, Valenzuela F, Astorga J, Fernandez A. Levels of the interleukins 17A, 22, and 23 and the S100 protein family in the gingival crevicular fluid of psoriatic patients with or without periodontitis. An Bras Dermatol. 2021 Mar-Apr;96(2):163-170. doi: 10.1016/j.abd.2020.08.008. Epub 2021 Jan 25. PMID 33531183